CLINICAL TRIAL: NCT02736955
Title: Open-Label Rollover Study for Continuing Valbenazine (NBI-98854) Administration for the Treatment of Tardive Dyskinesia
Brief Title: Rollover Study for Continuing Valbenazine (NBI-98854) Administration for the Treatment of Tardive Dyskinesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-1506
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

ARMS (1):
- Valbenazine (Experimental): Fixed dose of valbenazine administered once daily for up to 72 weeks
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine
  Other Names: NBI-98854

SUMMARY:
This Phase 3b, rollover study will provide participants who completed a Phase 3 valbenazine (NBI-98854) study open-label access to valbenazine (fixed doses administered once daily) for the treatment of adults with TD until valbenazine is anticipated to be available commercially or they complete 72 weeks of treatment. This study will allow enrollment of up to 150 medically stable male and female participants with TD who previously participated in and completed the NBI-98854-1304 (Kinect 3) or NBI-98854-1402 (Kinect 4) Phase 3 study.

DETAILED DESCRIPTION:
This study was terminated after 60 weeks due to the commercial availability of valbenazine.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in and completed the NBI-98854-1304 (Kinect 3) or NBI-98854-1402 (Kinect 4) Phase 3 study.
* Participants of childbearing potential must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently throughout the study and until 30 days after the last dose of valbenazine.
* If using maintenance medication(s) for schizophrenia or schizoaffective disorder, mood disorder, or other conditions, be on stable doses.
* Be in general good health.
* Have adequate hearing, vision, and language skills to perform the procedures specified in the protocol.

Exclusion Criteria:

* Have an active, clinically significant unstable medical condition within 1 month prior to screening.
* Have a known history of substance dependence, substance (drug) or alcohol abuse.
* Have a significant risk of suicidal or violent behavior.
* Have a known history of neuroleptic malignant syndrome.
* Have a known history of long QT syndrome or cardiac arrhythmia.
* Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed).
* Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than valbenazine) during the study.
* Have a blood loss ≥550 mL or donated blood within 30 days prior to Baseline.
* Have an allergy, hypersensitivity, or intolerance to tetrabenazine.
* Are currently pregnant or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Anaheim, California
  - National City, California
  - Norwalk, California
  - Oakland, California
  - San Bernardino, California
  - San Diego, California
  - Torrance, California
  - Hialeah, Florida
  - North Miami, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - Shreveport, Louisiana
  - Worcester, Massachusetts
  - Cedarhurst, New York
  - Dayton, Ohio
  - Shaker Heights, Ohio
  - Oklahoma City, Oklahoma
  - Norristown, Pennsylvania
  - Charleston, South Carolina
  - Franklin, Tennessee
  - Memphis, Tennessee
  - DeSoto, Texas
  - Fort Worth, Texas
  - Irving, Texas
  - Salt Lake City, Utah
  - Petersburg, Virginia
  - Spokane, Washington

REFERENCES:
- [Derived] Lindenmayer JP, Verghese C, Marder SR, Burke J, Jimenez R, Siegert S, Liang GS, O'Brien CF. A long-term, open-label study of valbenazine for tardive dyskinesia. CNS Spectr. 2021 Aug;26(4):345-353. doi: 10.1017/S109285292000108X. Epub 2020 May 18. PMID 32419679

RESULTS

PARTICIPANT FLOW:
Groups:
- Valbenazine 40 mg: Participants received 40 mg valbenazine oral capsule once daily for up to 60 weeks
- Valbenazine 80 mg: Participants received 40 mg valbenazine oral capsule once daily for 4 weeks, followed by 80 mg (provided as 2 x 40 mg valbenazine oral capsule) once daily for up to 56 weeks
- Valbenazine 40/80 mg: Participants received 40 mg valbenazine oral capsule once daily for 4 weeks. Participants were then increased to 80 mg (provided as 2 x 40 mg valbenazine oral capsule) once daily, and due to poor tolerance, were subsequently reduced back to one 40 mg valbenazine oral capsule once daily for the remainder of the study, up to 56 weeks
Period: Overall Study
Arm/Group | Valbenazine 40 mg | Valbenazine 80 mg | Valbenazine 40/80 mg
Started | 36 | 117 | 8
Completed | 29 | 103 | 6
Not Completed | 7 | 14 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valbenazine 40 mg | Valbenazine 80 mg | Valbenazine 40/80 mg | Total
Number analyzed (Participants) | 35 | 117 | 8 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (8.9) | 57.9 (8.8) | 59.3 (9.0) | 57.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 54 | 3 | 79
  Male | 13 | 63 | 5 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 52 | 1 | 57
  Not Hispanic or Latino | 31 | 65 | 7 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 14 | 30 | 3 | 47
  White | 21 | 86 | 4 | 111
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body Mass Index (BMI) at Baseline [Mean (Standard Deviation); unit: kg/m^2] | 29.15 (5.52) | 28.54 (5.48) | 30.55 (5.29) | 28.77 (5.46)
Primary Psychiatric Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia/schizoaffective disorder | 23 | 75 | 6 | 104
  Mood disorder | 12 | 42 | 2 | 56
Age at Diagnosis [Mean (Standard Deviation); unit: years] — Population: Age at diagnosis was not available for some participants.
  years
    Schizophrenia/Schizoaffective Disorder: number analyzed (Participants) | 18 | 72 | 6 | 96
    Schizophrenia/Schizoaffective Disorder | 27.1 (8.3) | 28.7 (11.4) | 25.3 (6.2) | 28.2 (10.6)
    Mood Disorder: number analyzed (Participants) | 11 | 42 | 2 | 55
    Mood Disorder | 36.0 (3.6) | 33.9 (2.1) | 46.0 (14.0) | 34.7 (1.8)
    Tardive Dyskinesia: number analyzed (Participants) | 25 | 91 | 8 | 124
    Tardive Dyskinesia | 48.3 (11.2) | 48.4 (9.5) | 43.8 (13.7) | 48.0 (10.1)
Scales [Mean (Standard Deviation); unit: units on a scale] — The Brief Psychiatric Rating Scale (BPRS) assesses the severity of psychopathology in patients with schizophrenia and other psychotic disorders by addressing 18 items. The severity of each item is rated on a scale of 1 (not present) to 7 (extremely severe) (total score range: 18 to 126). Higher scores represent greater symptom severity.
  The Clinical Global Impression of Tardive Dyskinesia-Severity (CGI-TD-severity) scale assesses the overall global severity of TD. The scale has 7 points from 1=normal, not at all ill to 7=among the most extremely ill patient. Population: Baseline CGI-TD-Severity Score is not available for one participant in the 80 mg valbenazine oral capsule treatment arm.
  units on a scale
    BPRS Score | 27.3 (6.3) | 26.1 (5.6) | 30.5 (9.2) | 26.6 (6.0)
    CGI-TD-Severity Score: number analyzed (Participants) | 35 | 116 | 8 | 159
    CGI-TD-Severity Score | 3.9 (1.1) | 3.9 (1.3) | 4.3 (0.7) | 3.9 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Monitored for Long-term Safety of Valbenazine
Description: Incidence of adverse events and monitoring of vital signs, clinical laboratory values, and electrocardiograms. All AEs were coded into preferred terms according to MedDRA (Medical Dictionary for Regulatory Activities) and classified by system organ class (SOC). Summaries of the incidence of all treatment-emergent AEs, treatment-related AEs, SAEs, and AEs leading to study drug discontinuation were prepared.
Time Frame: 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Valbenazine 40 mg | Valbenazine 80 mg | Valbenazine 40/80 mg
Number analyzed (Participants) | 35 | 117 | 8
Participants | 35 | 117 | 8

2. Secondary Outcome: Number of Participants With Clinical Response as Assessed by the Clinical Global Impression of Tardive Dyskinesia - Severity (CGI-TD-Severity) Scale
Description: Clinician's perspective of the participant's overall severity of TD symptoms. The CGI-TD-Severity is based on a 7-point scale (range: 1= "Normal, not at all ill" to 7= "Among the most extremely ill patient"). A clinical response was defined as a CGI-TD-S score equal to "1" or "2."
Time Frame: Baseline and Weeks 12, 24, 36, 48, and 60
Population: Safety analysis set: includes all participants who were enrolled in the study and received study drug, with the following two exclusions: (a) participants who withdrew from the study and returned all previously dispensed study drug with all doses present, and (b) participants who had no post-baseline data collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Valbenazine 40 mg | Valbenazine 80 mg | Valbenazine 40/80 mg
Number analyzed (Participants) | 35 | 117 | 8
Participants
  Baseline: number analyzed (Participants) | 35 | 116 | 8
  Baseline | 2 | 21 | 0
  Week 12: number analyzed (Participants) | 31 | 115 | 8
  Week 12 | 15 | 56 | 3
  Week 24: number analyzed (Participants) | 23 | 96 | 6
  Week 24 | 11 | 56 | 4
  Week 36: number analyzed (Participants) | 18 | 68 | 5
  Week 36 | 7 | 44 | 2
  Week 48: number analyzed (Participants) | 12 | 39 | 5
  Week 48 | 5 | 29 | 2
  Week 60: number analyzed (Participants) | 2 | 2 | 0
  Week 60 | 2 | 2 |

3. Secondary Outcome: Number of Participants With Clinical Response as Assessed by the Patient Satisfaction Questionnaire (PSQ)
Description: Participant's perspective of his/her satisfaction with valbenazine treatment. The PSQ is based on a 5-point scale (range: 1=very satisfied to 5=very dissatisfied). A clinical response was defined as a PSQ score equal to "1" or "2."
Time Frame: Baseline and Weeks 12, 24, 36, 48, and 60
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Valbenazine 40 mg | Valbenazine 80 mg | Valbenazine 40/80 mg
Number analyzed (Participants) | 35 | 117 | 8
Participants
  Baseline | 35 | 116 | 7
  Week 12: number analyzed (Participants) | 31 | 115 | 7
  Week 12 | 30 | 112 | 6
  Week 24: number analyzed (Participants) | 23 | 96 | 6
  Week 24 | 23 | 92 | 6
  Week 36: number analyzed (Participants) | 18 | 68 | 5
  Week 36 | 17 | 66 | 5
  Week 48: number analyzed (Participants) | 12 | 39 | 5
  Week 48 | 12 | 38 | 5
  Week 60: number analyzed (Participants) | 2 | 2 | 0
  Week 60 | 2 | 2 |

ADVERSE EVENTS:
Time Frame: Up to 60 weeks
Arm/Group | Valbenazine 40 mg | Valbenazine 80 mg | Valbenazine 40/80 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 3/117 | 1/8
Serious Adverse Events (participants affected / at risk) | 3/35 | 11/117 | 2/8
Other Adverse Events (participants affected / at risk) | 6/35 | 23/117 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine 40 mg (N=35) | Valbenazine 80 mg (N=117) | Valbenazine 40/80 mg (N=8)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Sepsis syndrome (Infections and infestations) | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine 40 mg (N=35) | Valbenazine 80 mg (N=117) | Valbenazine 40/80 mg (N=8)
Urinary tract infection (Infections and infestations) | 1 | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 4 | 0
Headache (Nervous system disorders) | 1 | 4 | 0
Tremor (Nervous system disorders) | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02736955/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT02736955/SAP_001.pdf